CLINICAL TRIAL: NCT04281602
Title: Biomarkers in Patients Suffering From Rheumatoid Arthritis Treated With Anti-interleukin-6 Therapy: a Prospective Monocentric Controlled Study
Brief Title: Biomarkers in Rheumatoid Arthritis Treated With Anti-interleukin-6 Therapy
Acronym: INTER-ACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01557-50
Record Dates: First submitted 2019-11-27; First posted 2020-02-24 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis patients: Adult patients suffering from rheumatoid arthritis, diagnosed according to American College of Rheumatology/European League Against Rheumatism 2010 criteria and requiring a anti-IL-6 treatment
- Healthy controls: Healthy controls not suffering from acute or chronic inflammatory disease at inclusion.

SUMMARY:
The use of anti-interleukin (IL)-6 therapy, including tocilizumab, in rheumatoid arthritis or giant cell arteritis, led to the improvement or even control of disease in some patients for whom no further therapeutic options were available. Nevertheless, the evaluation of the efficacy of these treatments are negatively impacted by the lack of reliable biomarkers. Indeed, usual inflammatory biomarkers used during the follow-up of these patients to detect persistent disease activity or intercurrent infection, such as C-reactive protein, fibrinogen and procalcitonin, are dependant on IL-6. Thse usual biomarkers cannot therefore be reliably used during anti-IL-6 therapy. Some other experimental biomarkers are totally or partially independent of IL-6, or even of inflammasome, and thus are credible candidates for the follow-up of patients treated with anti-IL-6 therapy.

Here investigators propose a controlled, prospective, monocentric, observational study evaluating several biomarkers, usual and experimental, in patients suffering from rheumatoid arthritis treated with anti-IL-6 therapy.

This study will include 25 patients suffering from rheumatoid arthritis requiring an anti-IL-6 therapy and 25 healthy controls.

In patients suffering from rheumatoid arthritis, usual and experimental biomarkers will be assessed at D0, D15, W24 and W52 from the introduction of anti-IL-6 therapy, or during an intercurrent infection.

Investigators thus hypothesized that experimental biomarker levels will still be increased at D15, contrary to usual biomarkers dependant on IL-6 which will be normal whereas rheumatoid arthritis is still active based on usual radiological and clinical criteria, and that all biomarkers will be normal a W24.

ELIGIBILITY:
Inclusion Criteria for patients:

* Adult patients suffering from rheumatoid arthritis diagnosed according to American College of Rheumatology/European League Against Rheumatism 2010 criteria and requiring an anti-IL-6 therapy by intravenous or subcutaneous injection
* Non-opposition of the patient

Inclusion Criteria for healthy controls:

* Adult patients not suffering from acute or chronic inflammatory disease at inclusion (normal C-reactive protein and fibrinogen levels)
* Non-opposition of the subject

Exclusion Criteria for patients:

* Patient is already treated with anti-IL-6 therapy
* Pregnancy or breastfeeding women
* Person under judicial protection, guardianship
* Patient suffering from another chronic inflammatory disease
* Patient suffering from another acute inflammatory disease at inclusion
* Person not beneficiaries of the social security system

Exclusion Criteria for healthy controls:

* Pregnancy or breastfeeding women
* Person under judicial protection, guardianship
* Patient suffering from acute or chronic inflammatory disease at inclusion
* Previous history of chronic inflammatory disease
* Ongoing anti-inflammatory or immunosuppressive treatment, except aspirin and derivatives at anti-platelet aggregation dose, non-steroidal anti-inflammatory drugs stopped for 10 days or systemic steroids stopped for 1 month
* Person not beneficiaries of the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and healthy controls followed at Caen, university hospital, in the department of rhumatology or internal medicine
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-01-02 (Estimated); Study Completion 2024-05-02 (Estimated)

PRIMARY OUTCOMES:
Levels of usual biomarkers (C-reactive protein, fibrinogen, procalcitonin, serum protein electrophoresis) | Day 15
  C-reactive protein and fibrinogen measured by turbidimetry; procalcitonin by an enzyme immunoassay kit, serum protein electrophoresis by electrophoresis
Levels of experimental biomarkers (IL-8, IL-1beta, IL-1RA, IL-4, IL-5, IL-6, IL-10, IL-12/23, IL-17, IL-18, IL-21, IFN-gamma, TNF-alpha, TGF-beta, S100 proteins, ceruloplasmin, C3, C4, CH50, serum amyloid A, factor VIII, neutrophil/lymphocyte ratio) | Day 15
  IL-8, IL-1beta, IL-1RA, IL-4, IL-5, IL-6, IL-10, IL-12/23, IL-17, IL-18, IL-21, IFN-gamma, TNF-alpha, TGF-beta and S100 proteins measured by Meso Scale Discovery assay, ceruloplasmin, C3, C4, serum amyloid A by nephelometry, CH50 by an enzyme immunoassay kit, factor VIII by turbidimetry, neutrophil/lymphocyte ratio by an automated method

SECONDARY OUTCOMES:
Levels of usual biomarkers (C-reactive protein, fibrinogen, procalcitonin, serum protein electrophoresis) | Day 15 compared to Day 0
  C-reactive protein and fibrinogen measured by turbidimetry; procalcitonin by an enzyme immunoassay kit, serum protein electrophoresis by electrophoresis
Levels of experimental biomarkers (IL-8, IL-1beta, IL-1RA, IL-4, IL-5, IL-6, IL-10, IL-12/23, IL-17, IL-18, IL-21, IFN-gamma, TNF-alpha, TGF-beta, S100 proteins, ceruloplasmin, C3, C4, CH50, serum amyloid A, factor VIII, neutrophil/lymphocyte ratio) | Day 15 compared to Day 0
  IL-8, IL-1beta, IL-1RA, IL-4, IL-5, IL-6, IL-10, IL-12/23, IL-17, IL-18, IL-21, IFN-gamma, TNF-alpha, TGF-beta and S100 proteins measured by Meso Scale Discovery assay, ceruloplasmin, C3, C4, serum amyloid A by nephelometry, CH50 by an enzyme immunoassay kit, factor VIII by turbidimetry, neutrophil/lymphocyte ratio by an automated method
Levels of usual biomarkers (C-reactive protein, fibrinogen, procalcitonin, serum protein electrophoresis, erythrocyte sedimentation rate) | Week 24 compared to Day 15
  C-reactive protein and fibrinogen measured by turbidimetry; procalcitonin by an enzyme immunoassay kit, serum protein electrophoresis by electrophoresis, erythrocyte sedimentation rate by an automated method
Levels of experimental biomarkers (IL-8, IL-1beta, IL-1RA, IL-4, IL-5, IL-6, IL-10, IL-12/23, IL-17, IL-18, IL-21, IFN-gamma, TNF-alpha, TGF-beta, S100 proteins, ceruloplasmin, C3, C4, CH50, serum amyloid A, factor VIII, neutrophil/lymphocyte ratio) | Week 24 compared to Day 15
  IL-8, IL-1beta, IL-1RA, IL-4, IL-5, IL-6, IL-10, IL-12/23, IL-17, IL-18, IL-21, IFN-gamma, TNF-alpha, TGF-beta and S100 proteins measured by Meso Scale Discovery assay, ceruloplasmin, C3, C4, serum amyloid A by nephelometry, CH50 by an enzyme immunoassay kit, factor VIII by turbidimetry, neutrophil/lymphocyte ratio by an automated method
Levels of usual biomarkers (C-reactive protein, fibrinogen, procalcitonin, serum protein electrophoresis, erythrocyte sedimentation rate) | Within 72 hours following infection occuring after week 24
  C-reactive protein and fibrinogen measured by turbidimetry; procalcitonin by an enzyme immunoassay kit, serum protein electrophoresis by electrophoresis, erythrocyte sedimentation rate by an automated method
Levels of experimental biomarkers (IL-8, IL-1beta, IL-1RA, IL-4, IL-5, IL-6, IL-10, IL-12/23, IL-17, IL-18, IL-21, IFN-gamma, TNF-alpha, TGF-beta, S100 proteins, ceruloplasmin, C3, C4, CH50, serum amyloid A, factor VIII, neutrophil/lymphocyte ratio) | Within 72 hours following infection occuring after week 24
  IL-8, IL-1beta, IL-1RA, IL-4, IL-5, IL-6, IL-10, IL-12/23, IL-17, IL-18, IL-21, IFN-gamma, TNF-alpha, TGF-beta and S100 proteins measured by Meso Scale Discovery assay, ceruloplasmin, C3, C4, serum amyloid A by nephelometry, CH50 by an enzyme immunoassay kit, factor VIII by turbidimetry, neutrophil/lymphocyte ratio by an automated method

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided